CLINICAL TRIAL: NCT03310619
Title: An Exploratory Phase 1/2 Trial To Evaluate The Safety And Efficacy Of JCAR017 Combinations In Subjects With Relapsed/Refractory B-Cell Malignancies (PLATFORM)
Brief Title: A Safety and Efficacy Trial of JCAR017 Combinations in Subjects With Relapsed/Refractory B-cell Malignancies
Acronym: PLATFORM
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JCAR017-BCM-002; U1111-1201-2046 (Registry Identifier: WHO)
Record Dates: First submitted 2017-09-25; First posted 2017-10-16 (Actual); Results first posted 2024-04-04 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-03

CONDITIONS: Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular
Keywords: JCAR017; B-Cell Malignancies; NHL; non-Hodgkin lymphoma; CAR T cells; chimeric antigen receptor; CC-220; Ibrutinib; relatlimab; nivolumab; CC-99282
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular | interventions — durvalumab; 3-(5-amino-2-methyl-4-oxoquinazolin-3(4H)-yl)piperidine-2,6-dione; ibrutinib; iberdomide; relatlimab; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Arm A: JCAR017 in combination with Durvalumab (Experimental): JCAR017 will be administered at a single flat dose of 50 x 10^6 CAR+T cells or 100 x 10^6 CAR+T cells. The combination agent will be administered at different doses and/ or schedules
  Interventions: Biological: JCAR017; Drug: Durvalumab
- Arm B: JCAR017 in combination with CC-122 (Experimental): This arm will test JCAR017 in combination with the CC-122. In adult subjects with R/R aggressive B-cell NHL. JCAR017 will be administered at a dose of 100 x 10^6 CAR+T cells. The combination agent will be administered at different doses
  Interventions: Biological: JCAR017; Drug: CC-122
- Arm C: JCAR017 in combination with CC-220 (Experimental): This arm will test JCAR017 in combination with CC-220. In adult subjects with R/R aggressive B-cell NHL. JCAR017 will be administered at a dose of 100 x 10^6 CAR+T cells. The combination agent will be administered at different doses
  Interventions: Biological: JCAR017; Drug: CC-220
- Arm D: JCAR017 in combination with Ibrutinib (Experimental): This arm will test JCAR017 in combination with ibrutinib. In adult subjects with R/R aggressive B-cell NHL. JCAR017 will be administered at a dose of 100 x 10^6 CAR+T cells. The combination agent will be administered at a fixed dose of 420 mg daily
  Interventions: Biological: JCAR017; Drug: Ibrutinib
- Arm E: JCAR017 in combination with relatlimab and/or nivolumab (Experimental): This arm will test JCAR017 in combination with relatlimab and/or nivolumab in adult subjects with R/R aggressive B-cell NHL. JCAR017 will be administered at a dose of 100 x 10^6 CAR+T cells. The combination agent will be administered at different doses and/or schedules
  Interventions: Biological: JCAR017; Drug: Relatlimab; Drug: Nivolumab
- Arm F: JCAR017 in combination with CC-99282 (Experimental): This arm will test JCAR017 in combination with CC-99282 in adult subjects with R/R aggressive B-cell NHL. JCAR017 will be administered at a dose of 100 x 10^6 CAR+T cells. The combination agent will be administered at different doses and/or schedules.
  Interventions: Biological: JCAR017; Drug: CC-99282

INTERVENTIONS:
Biological: JCAR017 — Gene modified autologous T cells
Drug: Durvalumab — Anti-PD-L1
  Other Names: MEDI4736
  Arms: Arm A: JCAR017 in combination with Durvalumab
Drug: CC-122 — Pleiotropic Pathway Modifier
  Arms: Arm B: JCAR017 in combination with CC-122
Drug: Ibrutinib — Ibrutinib
  Arms: Arm D: JCAR017 in combination with Ibrutinib
Drug: CC-220 — CC-220
  Arms: Arm C: JCAR017 in combination with CC-220
Drug: Relatlimab — Relatlimab
  Arms: Arm E: JCAR017 in combination with relatlimab and/or nivolumab
Drug: Nivolumab — Nivolumab
  Arms: Arm E: JCAR017 in combination with relatlimab and/or nivolumab
Drug: CC-99282 — CC-99282
  Arms: Arm F: JCAR017 in combination with CC-99282

SUMMARY:
This is a global, open-label, multi-arm, parallel multi-cohort, multi-center, Phase 1/2 study to determine the safety, tolerability, PK, efficacy and patient-reported quality of life of JCAR017 in combination with various agents. This protocol is intended to evaluate various drug combinations with JCAR017, as separate arms, over the life of the protocol, using the same objectives. Each combination will be evaluated separately (ie, the intention is not to compare between combinations) for the purposes of the objectives, trial design, and statistical analysis. The following combinations will be tested:

Arm A: JCAR017 in combination with durvalumab Arm B: JCAR017 in combination with CC-122 (avadomide) Arm C: JCAR017 in combination with CC-220 (iberdomide) Arm D: JCAR017 in combination with ibrutinib Arm E: JCAR017 in combination with relatlimab and/or nivolumab Arm F: JCAR017 in combination with CC-99282 Additional arms will be added by way of amendment once combination agents have been selected.

The study will consist of 2 parts: dose finding (Phase 1) and dose expansion (Phase 2). Dose expansion may occur in one or more arms.

DETAILED DESCRIPTION:
During Phase 1, different arms may be opened to test JCAR017 in combination with combination agent(s) in adult subjects with R/R aggressive B-cell NHL. Within each arm, different doses and schedules of JCAR017 and the combination agent(s) may be tested in several cohorts and subcohorts per arm. During Phase 2 of the study, the expansion of any dose level and schedule for any arm that has been shown to be safe may occur.

Arm A will test JCAR017 in combination with Durvalumab Arm B will test JCAR017 in combination with CC-122 Arm C will test JCAR017 in combination with CC-220 (iberdomide ) Arm D will test JCAR017 in combination with ibrutinib. Arm E will test JCAR017 in combination with relatlimab and/or nivolumab Arm F will test JCAR017 in combination with CC-99282 All subjects from Phase 1 and Phase 2 will be followed for 24 months following JCAR017 infusion. Post-study follow-up for survival, relapse, long-term toxicity (including new malignancies), and viral vector safety will continue under a separate long-term follow-up (LTFU) protocol for up to 15 years after the JCAR017 dose as per health authority regulatory guidelines.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is ≥ 18 years of age at the time of signing the informed consent form ().
2. Subject must understand and voluntarily sign an ICF prior to any study-related assessments/procedures being conducted.
3. Subject is willing and able to adhere to the study visit schedule and other protocol requirements.
4. Subject must have aggressive B-cell NHL according to "the 2016 revision of the WHO classification of lymphoid neoplasms", histologically confirmed at last relapse by the treating institution, defined as:

   1. Diffuse large B-cell lymphoma (DLBCL) Not otherwise specified (NOS) including transformed indolent Non-Hodgkin lymphoma (NHL)
   2. Follicular lymphoma Grade 3B
   3. T cell/histiocyte-rich large B-cell lymphoma
   4. Epstein-Barr virus (EBV) positive DLBCL, NOS
   5. Primary mediastinal (thymic) large B-cell lymphoma
   6. High grade B-cell lymphoma with MYC and BCL2 and/or BCL6 rearrangements with DLBCL histology (double/triple-hit lymphoma)
5. Subjects disease must have relapsed or be refractory to at least 2 prior lines of therapy. Previous therapy must have included a CD20-targeted agent and an anthracycline.
6. Subject must have

   1. Positron emission tomography (PET)-positive (Deauville score 4 or 5) and computed tomography (CT) measurable disease as per Lugano Classification
   2. Sum of product of perpendicular diameters (SPD) of up to 6 index lesions ≥ 25 cm2 by CT scan (not applicable to Arm A or B or subjects with Richter's transformation)
7. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1 at screening
8. Adequate organ function
9. Subjects must agree to not donate blood, organs, sperm or semen, and egg cells for usage in other individuals
10. Participants must agree to use effective contraception

Exclusion Criteria:

1. Subject has any significant medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from participating in the study based on investigator´s judgment.
2. Subject has any condition including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study based on investigator´s judgment.
3. Subject has any condition that confounds the ability to interpret data from the study based on investigator´s judgment.
4. Subjects with prior history of malignancies, other than aggressive R/R NHL, unless the subject has been free of the disease for ≥ 2 years with the exception of the following non-invasive malignancies:

   1. Basal cell carcinoma of the skin
   2. Squamous cell carcinoma of the skin
   3. Carcinoma in situ of the cervix
   4. Carcinoma in situ of the breast
   5. Incidental histologic finding of prostate cancer (T1a or T1b using the TNM [tumor, nodes, metastasis] clinical staging system) or prostate cancer that is curative.
   6. Other completely resected stage 1 solid tumor with low risk for recurrence
5. Prior treatment with any prior gene therap y product
6. Prior treatment with any adoptive T cell therapy; prior hematopoietic stem cell transplant (HSCT) is allowed
7. Allogeneic HSCT within 90 days of leukapheresis
8. Prior treatment with the combination agent from the assigned arm:

   1. Anti PD-1 or PD-L1 (Arm A and E)
   2. CC-122 (Arm B)
   3. CC-220 (Arm C)
   4. Prior treatment with ibrutinib is not exclusionary for subjects on any study arm
   5. Anti LAG-3 targeted agent (Arm E)
   6. CC-99282 (Arm F)
9. Presence of acute or chronic graft-versus-host disease (GVHD)
10. Presence of the following:

    1. Active hepatitis B or active hepatitis C infection
    2. History of or active human immunodeficiency virus (HIV) infection
11. Uncontrolled bacterial, viral or fungal infection at the time of leukapheresis, lymphodepleting chemotherapy or JCAR017 infusion
12. Any history of myocarditis (Arm E); history of any one of the following cardiovascular conditions within the past 6 months: Class III or IV heart failure as defined by the New York Heart Association (NYHA), cardiac angioplasty or stenting, myocardial infarction, unstable angina, or other clinically significant cardiac disease (all arms)
13. History or presence of clinically relevant central nervous system (CNS) pathology such as epilepsy, seizure, paresis, aphasia, stroke, severe brain injuries, dementia, Parkinson's disease, cerebellar disease, organic brain syndrome, or psychosis
14. Subjects with active CNS or cerebrospinal fluid (CSF) involvement by malignancy
15. Pregnant or nursing (lactating) women.
16. Subjects with active auto immune disorders/processes or active neurological or inflammatory disorders
17. For subjects to receive oral combination therapy (Arms B, C, D or F): History of a gastrointestinal (GI) condition or procedure that in the opinion of the investigator may affect oral drug absorption.
18. Progressive tumor invasion of venous or arterial vessels.
19. Deep venous thrombosis (DVT)/pulmonary embolism (PE) not managed on a stable regimen of anticoagulation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2017-12-20 (Actual); Primary Completion 2023-02-15 (Actual); Study Completion 2023-02-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (9):
- United States (9):
  - Local Institution - 011, Duarte, California
  - Local Institution - 022, Atlanta, Georgia
  - Local Institution - 014, Chicago, Illinois
  - Local Institution - 012, Boston, Massachusetts
  - Local Institution - 021, Boston, Massachusetts
  - Local Institution - 015, Omaha, Nebraska
  - Local Institution - 016, Philadelphia, Pennsylvania
  - Local Institution - 020, Pittsburgh, Pennsylvania
  - Local Institution - 013, Houston, Texas

REFERENCES:
- [Derived] Ernst M, Oeser A, Besiroglu B, Caro-Valenzuela J, Abd El Aziz M, Monsef I, Borchmann P, Estcourt LJ, Skoetz N, Goldkuhle M. Chimeric antigen receptor (CAR) T-cell therapy for people with relapsed or refractory diffuse large B-cell lymphoma. Cochrane Database Syst Rev. 2021 Sep 13;9(9):CD013365. doi: 10.1002/14651858.CD013365.pub2. PMID 34515338
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.BMSStudyConnect.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were only enrolled into the following groups:
  Arm A: Cohorts1 A and 1B, Arm B: Cohort 1A, Arm C: Cohort 1A, Arm D: Cohort 1A, Arm E: Cohort 1C, Arm F: Cohorts 1A and 1D.
Pre-assignment Details: Within each combination arm, up to 3 cohorts plus various sub cohorts (e.g., additional dose levels and schedules) may be tested. Data was pre-determined to be collected and reported combined as specified per arm and not per cohort.
Groups:
- Arm A: Cohort 1A JCAR017 Plus Durvalumab (Post-JCAR017 Infusion): JCAR017 was administered at a dose of (50 x 10^6 CAR+ T cells). On Day 29 after infusion, Durvalumab was administered at a low dose. On day 43 after infusion Durvalumab was administered at a mid-dose and on days 57 and 85 after infusion was administered at a high dose. Participants who reached a partial response 3 months after JCAR017 infusion could continue Durvalumab until progression for a maximum total duration of 12 months.
- Arm A: Cohort 1B JCAR017 Plus Durvalumab (Post-JCAR017 Infusion): JCAR017 was administered at a dose of (100 x 10^6 CAR+ T cells). On Day 29 after infusion, Durvalumab was administered at a low dose. On day 43 after infusion Durvalumab was administered at a mid-dose and on days 57 and 85 after infusion was administered at a high dose. Participants who reached a partial response 3 months after JCAR017 infusion could continue Durvalumab until progression for a maximum total duration of 12 months.
- Arm B: Cohort 1A JCAR017 Plus CC-122 (Post-JCAR017 Infusion): JCAR017 was administered at a dose of 100 x 10^6 CAR+T cells. Between days 29 and 180 after infusion participants received a standard dose of CC-122, 5 out of 7 days. Participants who reached a partial response or stable disease 6 months (Day 180) after JCAR017 infusion could continue CC-122 until progression or for up to Month 24, whatever was earlier.
- Arm C: Cohort 1A JCAR017 Plus CC-220 (Iberdomide) (Post-JCAR017 Infusion): JCAR017 was administered at a dose of 100 x 10^6 CAR+T cells. Between Days 15 -21 post infusion, CC-220 was administered at a standard dose. Participants who reached a partial response or stable disease at Day 85 (Month 3) after JCAR017 infusion could continue CC-220 until progression or for up to Month 12, whichever was earlier.
- Arm D: Cohort 1A JCAR017 Plus Ibrutinib (Pre- and Post-JCAR017 Infusion): Ibrutinib was administered from 35 days before to 85 days post JCAR017 infusion which was administered at a dose of 100 x 10^6 CAR+T cells. Participants received ibrutinib until 85 days post-infusion (Month 3).
- Arm E: Cohort 1C JCAR017 Plus Relatlimab and/or Nivolumab (Post-JCAR017 Infusion): JCAR017 was administered at a dose of 100 x 10^6 CAR+T cells. On days 8, 22, 36 post infusion, nivolumab was administered at a low dose. On days 57 and 85 post infusion, participants received nivolumab at a higher dose. Participants received nivolumab until Day 85 (Month 3).
- Arm F: Cohort 1A Cohort 1A and 1D JCAR017 Plus CC-99282 (Post-JCAR017 Infusion): JCAR017 was administered at a dose of (100 x 10^6 CAR+ T cells). Starting on Day 8 post infusion, CC-99282 was administered every 7 days. Participants received CC-99282 until Day 85 (Month 3)
- Arm F: Cohort 1D Cohort 1A and 1D JCAR017 Plus CC-99282 (Post-JCAR017 Infusion): JCAR017 was administered at a dose of (100 x 10^6 CAR+ T cells). Starting on Day 1 post infusion, CC-99282 was administered every 7 days. Participants received CC-99282 until Day 85 (Month 3)
Period: Pre-Treatment Period
Arm/Group | Arm A: Cohort 1A JCAR017 Plus Durvalumab (Post-JCAR017 Infusion) | Arm A: Cohort 1B JCAR017 Plus Durvalumab (Post-JCAR017 Infusion) | Arm B: Cohort 1A JCAR017 Plus CC-122 (Post-JCAR017 Infusion) | Arm C: Cohort 1A JCAR017 Plus CC-220 (Iberdomide) (Post-JCAR017 Infusion) | Arm D: Cohort 1A JCAR017 Plus Ibrutinib (Pre- and Post-JCAR017 Infusion) | Arm E: Cohort 1C JCAR017 Plus Relatlimab and/or Nivolumab (Post-JCAR017 Infusion) | Arm F: Cohort 1A Cohort 1A and 1D JCAR017 Plus CC-99282 (Post-JCAR017 Infusion) | Arm F: Cohort 1D Cohort 1A and 1D JCAR017 Plus CC-99282 (Post-JCAR017 Infusion)
Started (Started = Leukopheresed) | 11 | 9 | 13 | 1 | 17 | 2 | 7 | 2
Completed | 8 | 8 | 11 | 1 | 16 | 2 | 5 | 2
Not Completed | 3 | 1 | 2 | 0 | 1 | 0 | 2 | 0
Not completed — Death | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Other reasons | 2 | 1 | 2 | 0 | 0 | 0 | 2 | 0
Period: Treatment Period
Arm/Group | Arm A: Cohort 1A JCAR017 Plus Durvalumab (Post-JCAR017 Infusion) | Arm A: Cohort 1B JCAR017 Plus Durvalumab (Post-JCAR017 Infusion) | Arm B: Cohort 1A JCAR017 Plus CC-122 (Post-JCAR017 Infusion) | Arm C: Cohort 1A JCAR017 Plus CC-220 (Iberdomide) (Post-JCAR017 Infusion) | Arm D: Cohort 1A JCAR017 Plus Ibrutinib (Pre- and Post-JCAR017 Infusion) | Arm E: Cohort 1C JCAR017 Plus Relatlimab and/or Nivolumab (Post-JCAR017 Infusion) | Arm F: Cohort 1A Cohort 1A and 1D JCAR017 Plus CC-99282 (Post-JCAR017 Infusion) | Arm F: Cohort 1D Cohort 1A and 1D JCAR017 Plus CC-99282 (Post-JCAR017 Infusion)
Started (Started = entered treatment period) | 8 | 8 | 11 | 1 | 16 | 2 | 5 | 2
Safety Set (Received a dose of JCAR017 Cell Product or at least one dose of the combination agent.) | 8 | 8 | 11 | 1 | 17 (1 Participant who died in pre-treatment period received Ibrutinib prior to entering the treatment period and was thus included in the safety set.) | 2 | 4 | 2
Completed | 6 | 5 | 4 | 0 | 12 | 2 | 3 | 0
Not Completed | 2 | 3 | 7 | 1 | 4 | 0 | 2 | 2
Not completed — Death | 1 | 2 | 0 | 0 | 1 | 0 | 2 | 0
Not completed — Adverse Event | 0 | 1 | 4 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by participant | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Study terminated by sponsor | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0
Not completed — Other reasons | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: Cohort 1A JCAR017 Plus Durvalumab (Post-JCAR017 Infusion) | Arm A: Cohort 1B JCAR017 Plus Durvalumab (Post-JCAR017 Infusion) | Arm B: Cohort 1A JCAR017 Plus CC-122 (Post-JCAR017 Infusion) | Arm C: Cohort 1A JCAR017 Plus CC-220 (Iberdomide) (Post-JCAR017 Infusion) | Arm D: Cohort 1A JCAR017 Plus Ibrutinib (Pre- and Post-JCAR017 Infusion) | Arm E: Cohort 1C JCAR017 Plus Relatlimab and/or Nivolumab (Post-JCAR017 Infusion) | Arm F: Cohort 1A Cohort 1A and 1D JCAR017 Plus CC-99282 (Post-JCAR017 Infusion) | Arm F: Cohort 1D Cohort 1A and 1D JCAR017 Plus CC-99282 (Post-JCAR017 Infusion) | Total
Number analyzed (Participants) | 11 | 9 | 13 | 1 | 17 | 2 | 7 | 2 | 62
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.9 (8.40) | 68.6 (6.65) | 60.8 (14.66) | 69.0 (NA) — Insufficient number of participants to calculate SD. | 56.5 (12.19) | 66.5 (2.12) | 66.6 (14.14) | 55.0 (19.8) | 61.7 (11.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 1 | 0 | 7 | 0 | 4 | 1 | 19
  Male | 8 | 6 | 12 | 1 | 10 | 2 | 3 | 1 | 43
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 0 | 0 | 2 | 0 | 1 | 0 | 5
  Not Hispanic or Latino | 10 | 8 | 13 | 1 | 15 | 2 | 6 | 2 | 57
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: Participants] — Population: Race
  Participants
    AMERICAN INDIAN OR ALASKA NATIVE | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
    ASIAN | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 3
    BLACK OR AFRICAN AMERICAN | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 3
    WHITE | 9 | 9 | 12 | 1 | 11 | 2 | 6 | 1 | 51
    OTHER | 1 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose-Limiting Toxicity (DLT)
Description: Participants enrolled in Phase 1 are considered evaluable for DLTs if they received an infusion of conforming JCAR017 cell product and at least one dose of the combination agent and completed the specified DLT evaluation period or if they have received an infusion of conforming JCAR017 cell product and at least one dose of the combination agent and experience a DLT during the DLT evaluation period.
Time Frame: From first dose of the combination agent until 1 month (28 days) after JCAR017 infusion (pre- JCAR017 cohort) or from JCAR017 infusion until 1 month (28 days) after the first dose of combination agent (post-JCAR017 cohort)
Population: Dose-Limiting Toxicity Evaluable Participants. Prespecified to be reported per Arm and not per cohort.
Measure: Count of Participants; unit: Participants
Groups:
- Arm A: Cohort 1A and 1B JCAR017 Plus Durvalumab (Post-JCAR017 Infusion): JCAR017 was administered at a dose of 50 x 10^6 CAR+T cells (dose level 1 [DL1]) or 100 x 10^6 CAR+T cells (DL2). On Day 29 after infusion, Durvalumab was administered at different doses and/ or schedules. Participants from both phases and all cohorts who reached a partial response 3 months after JCAR017 infusion could continue durvalumab until progression for a maximum total duration of 12 months.
- Arm B: JCAR017 Plus CC-122 (Post-JCAR017 Infusion): JCAR017 was administered at a dose of 100 x 10^6 CAR+T cells (DL2). On Day 29 after infusion, CC-122 was administered at different doses. Participants who reach a partial response or stable disease 6 months (Day 180) after JCAR017 infusion could continue CC-122 until progression or for up to Month 24, whatever was earlier.
- Arm C: JCAR017 Plus CC-220 (Iberdomide) (Post-JCAR017 Infusion): JCAR017 was administered at a dose of 100 x 10^6 CAR+T cells (DL2). Between Days 1 -21 post infusion, CC-220 was administered at different doses and/or schedules. Participants who reached a partial response or stable disease at Day 85 (Month 3) after JCAR017 infusion could continue CC-220 until progression or for up to Month 12, whichever was earlier.
- Arm D: JCAR017 Plus Ibrutinib (Pre- and Post-JCAR017 Infusion): Ibrutinib was administered at different doses on Day 1. On day 35, JCAR017 was administered at a dose of 100 x 10^6 CAR+T cells (DL2), followed again by Ibrutinib at different doses. Participants received ibrutinib until 85 days post-infusion (Month 3).
- Arm E: JCAR017 Plus Relatlimab and/or Nivolumab (Post-JCAR017 Infusion): JCAR017 was administered at a dose of 100 x 10^6 CAR+T cells (DL2). On day 8 or day 15 post infusion, relatlimab and nivolumab were administered at different doses and/or schedules. Participants received relatlimab and/or nivolumab until Day 85 (Month 3).
- Arm F: Cohort 1A and 1D JCAR017 Plus CC-99282 (Post-JCAR017 Infusion): JCAR017 was administered at a dose of 100 x 10^6 CAR+T cells (DL2). On day 1, 8, or day 15 post infusion CC-99282 was administered at different doses and/or schedules. Participants received CC-99282 until Day 85 (Month 3).
Arm/Group | Arm A: Cohort 1A and 1B JCAR017 Plus Durvalumab (Post-JCAR017 Infusion) | Arm B: JCAR017 Plus CC-122 (Post-JCAR017 Infusion) | Arm C: JCAR017 Plus CC-220 (Iberdomide) (Post-JCAR017 Infusion) | Arm D: JCAR017 Plus Ibrutinib (Pre- and Post-JCAR017 Infusion) | Arm E: JCAR017 Plus Relatlimab and/or Nivolumab (Post-JCAR017 Infusion) | Arm F: Cohort 1A and 1D JCAR017 Plus CC-99282 (Post-JCAR017 Infusion)
Number analyzed (Participants) | 14 | 8 | 1 | 8 | 2 | 5
Participants | 0 | 2 | 1 | 1 | 0 | 0

2. Primary Outcome: Complete Response Rate (CRR)
Description: Percentage of participants achieving a complete response (CR). CR is complete radiologic response (CRR) and complete metabolic response (CMR). CR was measured using CT and PET and assessed for the presence of index and non-index lesions, spleen size, and the absence of new lesions or diseased bone marrow.
  To be considered as having CRR participants had to have all of the following:
  * Index lesions - longest transverse diameter of nodal lesions ≤ 1.5 cm and the absence of extranodal disease.
  * Non-index lesions - the absence of non-index lesions.
  * Spleen size <13 cm
  * The absence of new lesions
  * Normal bone marrow assessment
  To be considered as having CMR participants had to have all of the following:
  * A score of 1, 2, or 3 with or without residual mass on 5-PS for index and non-index lesions.
  * The absence of new lesions
  * No evidence of FDG-avid disease in marrow and a normal bone marrow assessment
Time Frame: At 3 and 6 months post-JCAR017 infusion.
Population: All participants in the combination treated set. The combination treated set included all participants who received an infusion of conforming JCAR017 cell product and at least one dose of the combination agent. Prespecified to be reported per Arm and not per cohort.
Measure: Number (95% Confidence Interval); unit: Percent of Participants
Groups:
- Arm A: JCAR017 Plus Durvalumab (Post-JCAR017 Infusion): JCAR017 was administered at a dose of 50 x 10^6 CAR+T cells (dose level 1 [DL1]) or 100 x 10^6 CAR+T cells (DL2). On Day 29 after infusion, Durvalumab was administered at different doses and/ or schedules. Participants from both phases and all cohorts who reached a partial response 3 months after JCAR017 infusion could continue durvalumab until progression for a maximum total duration of 12 months.
- Arm B: Cohort 1A: JCAR017 was administered at a dose of 100 x 10^6 CAR+T cells (DL2). On Day 29 after infusion, CC-122 was administered at different doses. Participants who reach a partial response or stable disease 6 months (Day 180) after JCAR017 infusion could continue CC-122 until progression or for up to Month 24, whatever was earlier.
- Arm F: JCAR017 Plus CC-99282 (Post-JCAR017 Infusion): JCAR017 was administered at a dose of 100 x 10^6 CAR+T cells (DL2). On day 1, 8, or day 15 post infusion CC-99282 was administered at different doses and/or schedules. Participants received CC-99282 until Day 85 (Month 3).
Arm/Group | Arm A: JCAR017 Plus Durvalumab (Post-JCAR017 Infusion) | Arm B: Cohort 1A | Arm C: JCAR017 Plus CC-220 (Iberdomide) (Post-JCAR017 Infusion) | Arm D: JCAR017 Plus Ibrutinib (Pre- and Post-JCAR017 Infusion) | Arm E: JCAR017 Plus Relatlimab and/or Nivolumab (Post-JCAR017 Infusion) | Arm F: JCAR017 Plus CC-99282 (Post-JCAR017 Infusion)
Number analyzed (Participants) | 14 | 8 | 1 | 15 | 2 | 5
Percent of Participants
  CRR at 3 Months | 71.4 [41.9 to 91.6] | 62.5 [24.5 to 91.5] | 0.0 [0.0 to 97.5] | 46.7 [21.3 to 73.4] | 0.0 [0.0 to 84.2] | 60.0 [14.7 to 94.7]
  CRR at 6 Months | 78.6 [49.2 to 95.3] | 62.5 [24.5 to 91.5] | 0.0 [0.0 to 97.5] | 53.3 [26.6 to 78.7] | 0.0 [0.0 to 84.2] | 60.0 [14.7 to 94.7]

3. Secondary Outcome: European Organisation for Research and Treatment of Cancer - Quality of Life C30 Questionnaire (EORTC QLQ-C30) Scores - Phase 2
Description: The EORTC QLQ-C30 is composed of five functional scales (physical, role, emotional, cognitive and social), three symptom scales (fatigue, nausea/vomiting, and pain), a global health status/health-related quality of life (HRQoL) scale, and six single items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties). The questionnaire is scored on a 4-point Likert response scale: 1 = not at all, 2 = a little, 3 = quite a bit, and 4 = very much.
  The raw score is calculated as the average of the items that contribute to the scale. The final scores are calculated via linear transformation of raw scores and range from 0 to 100.
  For functional scales (physical, role, emotional, social, cognitive and global health) higher scores indicate better QoL.
  For symptom scales (fatigue, nausea and vomiting and pain) and single items (dyspnea, insomnia, appetite loss, constipation, diarrhea and financial difficulties) lower scores indicate fewer symptoms, i.e. better QoL.
Time Frame: At baseline and 29 days and 57 days post JCAR017 dose
Population: All participants in the combination treated set with baseline or on treatment HRQoL Scores. The combination treated set included all participants who received an infusion of conforming JCAR017 cell product and at least one dose of the combination agent. Data was not, nor will ever be collected for Arms C, D, E, and F since participants in these arms did not enter phase 2. Prespecified to be reported per Arm and not per cohort.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Arm A: JCAR017 Plus Durvalumab (Post-JCAR017 Infusion) | Arm B: Cohort 1A | Arm C: JCAR017 Plus CC-220 (Iberdomide) (Post-JCAR017 Infusion) | Arm D: JCAR017 Plus Ibrutinib (Pre- and Post-JCAR017 Infusion) | Arm E: JCAR017 Plus Relatlimab and/or Nivolumab (Post-JCAR017 Infusion) | Arm F: JCAR017 Plus CC-99282 (Post-JCAR017 Infusion)
Number analyzed (Participants) | 14 | 7 | 0 | 0 | 0 | 0
Score on a scale
  Global Health Status - Baseline: number analyzed (Participants) | 12 | 7 | 0 | 0 | 0 | 0
  Global Health Status - Baseline | 72.92 (20.140) | 80.95 (16.467) |  |  |  |
  Global Health Status - JCAR017 Day 29 | 70.24 (12.957) | 85.71 (20.813) |  |  |  |
  Global Health Status - JCAR017 Day 57 | 75.60 (13.660) | 89.29 (12.467) |  |  |  |
  Physical Functioning - Baseline: number analyzed (Participants) | 12 | 7 | 0 | 0 | 0 | 0
  Physical Functioning - Baseline | 80.00 (23.613) | 86.67 (13.333) |  |  |  |
  Physical Functioning - JCAR017 Day 29 | 80.48 (22.716) | 91.43 (10.690) |  |  |  |
  Physical Functioning - JCAR017 Day 57 | 81.90 (22.710) | 87.62 (15.119) |  |  |  |
  Role Functioning - Baseline: number analyzed (Participants) | 12 | 7 | 0 | 0 | 0 | 0
  Role Functioning - Baseline | 68.06 (35.858) | 78.57 (28.406) |  |  |  |
  Role Functioning - JCAR017 Day 29 | 75.00 (30.487) | 88.10 (18.545) |  |  |  |
  Role Functioning - JCAR017 Day 57 | 77.38 (27.431) | 83.33 (25.459) |  |  |  |
  Emotional Functioning - Baseline: number analyzed (Participants) | 12 | 7 | 0 | 0 | 0 | 0
  Emotional Functioning - Baseline | 77.08 (21.059) | 85.71 (12.467) |  |  |  |
  Emotional Functioning -JCAR017 Day 29 | 86.90 (16.894) | 91.67 (12.729) |  |  |  |
  Emotional Functioning - JCAR017 Day 57 | 85.71 (16.803) | 89.29 (10.446) |  |  |  |
  Cognitive Functioning - Baseline: number analyzed (Participants) | 12 | 7 | 0 | 0 | 0 | 0
  Cognitive Functioning - Baseline | 81.94 (18.060) | 95.24 (8.133) |  |  |  |
  Cognitive Functioning - JCAR017 Day 29 | 88.10 (13.757) | 92.86 (13.113) |  |  |  |
  Cognitive Functioning - JCAR017 Day 57 | 94.05 (12.416) | 92.86 (13.113) |  |  |  |
  Social Functioning - Baseline: number analyzed (Participants) | 12 | 7 | 0 | 0 | 0 | 0
  Social Functioning - Baseline | 69.44 (36.121) | 76.19 (23.288) |  |  |  |
  Social Functioning - JCAR017 Day 29 | 69.05 (21.540) | 88.10 (15.853) |  |  |  |
  Social Functioning - JCAR017 Day 57 | 80.95 (20.524) | 85.71 (20.250) |  |  |  |
  Fatigue - Baseline: number analyzed (Participants) | 12 | 7 | 0 | 0 | 0 | 0
  Fatigue - Baseline | 37.96 (30.506) | 14.29 (16.623) |  |  |  |
  Fatigue - JCAR017 Day 29 | 26.98 (18.853) | 23.81 (18.624) |  |  |  |
  Fatigue - JCAR017 Day 57 | 32.54 (19.715) | 22.22 (22.222) |  |  |  |
  Nausea and Vomiting - Baseline: number analyzed (Participants) | 12 | 7 | 0 | 0 | 0 | 0
  Nausea and Vomiting - Baseline | 11.11 (28.721) | 7.14 (13.113) |  |  |  |
  Nausea and Vomiting - JCAR017 Day 29 | 9.52 (15.627) | 7.14 (8.909) |  |  |  |
  Nausea and Vomiting - JCAR017 Day 57 | 9.52 (14.194) | 0.00 (0.00) |  |  |  |
  Pain - Baseline: number analyzed (Participants) | 12 | 7 | 0 | 0 | 0 | 0
  Pain - Baseline | 34.72 (35.146) | 16.67 (19.245) |  |  |  |
  Pain - JCAR017 Day 29 | 20.24 (29.365) | 16.67 (19.245) |  |  |  |
  Pain - JCAR017 Day 57 | 22.62 (30.387) | 14.29 (20.250) |  |  |  |
  Dyspnea - Baseline: number analyzed (Participants) | 12 | 7 | 0 | 0 | 0 | 0
  Dyspnea - Baseline | 16.67 (17.408) | 4.76 (12.599) |  |  |  |
  Dyspnea - JCAR017 Day 29 | 21.43 (21.111) | 4.76 (12.599) |  |  |  |
  Dyspnea - JCAR017 Day 57 | 14.29 (17.118) | 4.76 (12.599) |  |  |  |
  Insomnia - Baseline: number analyzed (Participants) | 12 | 7 | 0 | 0 | 0 | 0
  Insomnia - Baseline | 41.67 (35.176) | 23.81 (25.198) |  |  |  |
  Insomnia - JCAR017 Day 29 | 16.67 (28.495) | 19.05 (14.29) |  |  |  |
  Insomnia - JCAR017 Day 57 | 35.71 (33.242) | 19.05 (17.817) |  |  |  |
  Appetite Loss - Baseline: number analyzed (Participants) | 12 | 7 | 0 | 0 | 0 | 0
  Appetite Loss - Baseline | 25.00 (32.177) | 14.29 (17.817) |  |  |  |
  Appetite Loss - JCAR017 Day 29 | 26.19 (26.726) | 9.52 (16.265) |  |  |  |
  Appetite Loss - JCAR017 Day 57 | 21.43 (28.063) | 4.76 (12.599) |  |  |  |
  Constipation - Baseline: number analyzed (Participants) | 12 | 7 | 0 | 0 | 0 | 0
  Constipation - Baseline | 13.89 (30.011) | 4.76 (12.599) |  |  |  |
  Constipation - JCAR017 Day 29 | 11.90 (28.063) | 4.76 (12.599) |  |  |  |
  Constipation - JCAR017 Day 57 | 14.29 (17.118) | 0.00 (0.000) |  |  |  |
  Diarrhea - Baseline: number analyzed (Participants) | 12 | 7 | 0 | 0 | 0 | 0
  Diarrhea - Baseline | 5.56 (12.975) | 9.52 (16.265) |  |  |  |
  Diarrhea - JCAR017 Day 29 | 7.14 (14.194) | 4.76 (12.599) |  |  |  |
  Diarrhea - JCAR017 Day 57 | 0.00 (0.000) | 9.52 (16.265) |  |  |  |
  Financial Difficulties - Baseline: number analyzed (Participants) | 12 | 7 | 0 | 0 | 0 | 0
  Financial Difficulties - Baseline | 30.56 (36.121) | 28.57 (29.991) |  |  |  |
  Financial Difficulties - JCAR017 Day 29 | 19.05 (31.254) | 23.81 (31.706) |  |  |  |
  Financial Difficulties - JCAR017 Day 57 | 21.43 (30.959) | 28.57 (29.991) |  |  |  |

4. Secondary Outcome: EuroQol- 5 Dimensions of Health Visual Analogue Scale (EQ-5D VAS) Scores - Phase 2
Description: The EuroQol- 5 Dimensions of Health Visual Analogue Scale (EQ-5D VAS) records the participant's self-rated health on a vertical visual analogue scale, where the endpoints are scored from 0 to 100 i.e., 'The worst health you can imagine' (score of 0) to 'The best health you can imagine' (score of 100). Higher scores indicate better health outcomes.
Time Frame: At baseline and 1, 29, 57, 85, 180, 270, 365, 545, and 730 days post JCAR017 dose
Population: All participants in the combination treated set with baseline or on treatment HRQoL Scores. The combination treated set included all participants who received an infusion of conforming JCAR017 cell product and at least one dose of the combination agent. Data was not, nor will ever be collected for Arms C, D, E, and F as participants in these Arms did not enter phase 2. Prespecified to be reported per Arm and not per cohort.
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Arm A: JCAR017 Plus Durvalumab (Post-JCAR017 Infusion) | Arm B: Cohort 1A | Arm C: JCAR017 Plus CC-220 (Iberdomide) (Post-JCAR017 Infusion) | Arm D: JCAR017 Plus Ibrutinib (Pre- and Post-JCAR017 Infusion) | Arm E: JCAR017 Plus Relatlimab and/or Nivolumab (Post-JCAR017 Infusion) | Arm F: JCAR017 Plus CC-99282 (Post-JCAR017 Infusion)
Number analyzed (Participants) | 14 | 7 | 0 | 0 | 0 | 0
Score on a Scale
  Baseline: number analyzed (Participants) | 13 | 7 | 0 | 0 | 0 | 0
  Baseline | 69.5 (21.83) | 82.6 (12.31) |  |  |  |
  JCAR017 Day 1 | 75.1 (13.62) | 89.1 (12.13) |  |  |  |
  JCAR017 Day 29 | 77.5 (18.93) | 90.9 (10.33) |  |  |  |
  JCAR017 Day 57 | 81.2 (16.20) | 90.3 (9.43) |  |  |  |
  JCAR017 Day 85: number analyzed (Participants) | 10 | 6 | 0 | 0 | 0 | 0
  JCAR017 Day 85 | 88.4 (8.47) | 93.0 (4.98) |  |  |  |
  JCAR017 Day 180: number analyzed (Participants) | 7 | 4 | 0 | 0 | 0 | 0
  JCAR017 Day 180 | 86.0 (10.68) | 90.8 (13.96) |  |  |  |
  Follow-up - Day 270: number analyzed (Participants) | 6 | 2 | 0 | 0 | 0 | 0
  Follow-up - Day 270 | 88.7 (7.50) | 96.0 (1.41) |  |  |  |
  Follow-up - Day 365: number analyzed (Participants) | 5 | 2 | 0 | 0 | 0 | 0
  Follow-up - Day 365 | 89.2 (15.22) | 98.0 (2.83) |  |  |  |
  Follow-up - Day 545: number analyzed (Participants) | 3 | 1 | 0 | 0 | 0 | 0
  Follow-up - Day 545 | 89.7 (0.58) | 95.0 (NA) — Insufficient number of participants to calculate SD. |  |  |  |
  Follow-up - Day 730/EOS: number analyzed (Participants) | 4 | 3 | 0 | 0 | 0 | 0
  Follow-up - Day 730/EOS | 79.3 (15.84) | 96.3 (3.21) |  |  |  |

5. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: An AE is any noxious, unintended, or untoward medical occurrence that may appear or worsen in a participant during the course of a study. It may be a new intercurrent illness, a worsening concomitant illness, an injury, or any concomitant impairment of the participant's health, including laboratory test values, regardless of etiology. Any worsening (i.e., any clinically significant adverse change in the frequency or intensity of a preexisting condition) is also considered an AE. All participants were monitored for AEs during the study. Assessments included monitoring of any or all of the following parameters: the participant's clinical symptoms, laboratory, pathological, radiological or surgical findings, physical examination findings, or findings from other tests and/or procedures.
Time Frame: Up to 3 months after the dose of JCAR017 or after the last dose of the combination agent, whichever occurred last (an average of 6.5 months up until a max of 9.5 months)
Population: Safety Set - All participants who received an infusion of conforming JCAR017 cell product or at least one dose of the combination agent. Prespecified to be reported per Arm and not per cohort.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: JCAR017 Plus Durvalumab (Post-JCAR017 Infusion) | Arm B: Cohort 1A | Arm C: JCAR017 Plus CC-220 (Iberdomide) (Post-JCAR017 Infusion) | Arm D: JCAR017 Plus Ibrutinib (Pre- and Post-JCAR017 Infusion) | Arm E: JCAR017 Plus Relatlimab and/or Nivolumab (Post-JCAR017 Infusion) | Arm F: JCAR017 Plus CC-99282 (Post-JCAR017 Infusion)
Number analyzed (Participants) | 16 | 11 | 1 | 17 | 2 | 6
Participants | 16 | 11 | 1 | 17 | 2 | 6

6. Secondary Outcome: Number of Participants With Severe Adverse Events (SAEs)
Description: An SAE is any AE occurring at any dose that:
  * Results in death;
  * Is life-threatening (i.e., in the opinion of the Investigator, the participant is at immediate risk of death from the AE);
  * Requires inpatient hospitalization or prolongation of existing hospitalization (hospitalization is defined as an inpatient admission, regardless of length of stay);
  * Results in persistent or significant disability/incapacity (a substantial disruption of the participant's ability to conduct normal life functions);
  * Is a congenital anomaly/birth defect;
  * Constitutes an important medical event.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: JCAR017 Plus Durvalumab (Post-JCAR017 Infusion) | Arm B: Cohort 1A | Arm C: JCAR017 Plus CC-220 (Iberdomide) (Post-JCAR017 Infusion) | Arm D: JCAR017 Plus Ibrutinib (Pre- and Post-JCAR017 Infusion) | Arm E: JCAR017 Plus Relatlimab and/or Nivolumab (Post-JCAR017 Infusion) | Arm F: JCAR017 Plus CC-99282 (Post-JCAR017 Infusion)
Number analyzed (Participants) | 16 | 11 | 1 | 17 | 2 | 6
Participants | 10 | 7 | 1 | 6 | 2 | 3

7. Secondary Outcome: Change From Baseline in White Blood Cell and Platelet Numbers
Description: White blood cell, and platelet counts. Baseline is defined as the last measurement on or prior to any study treatment.
Time Frame: 85 days after the dose of JCAR017 for Arms A, B, D, E, and F; 57 days after the dose of JCAR017 for Arm C
Population: All treated participants with baseline and Day 85/Day 57 hematology laboratory values. Prespecified to be reported per Arm and not per cohort.
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | Arm A: JCAR017 Plus Durvalumab (Post-JCAR017 Infusion) | Arm B: Cohort 1A | Arm C: JCAR017 Plus CC-220 (Iberdomide) (Post-JCAR017 Infusion) | Arm D: JCAR017 Plus Ibrutinib (Pre- and Post-JCAR017 Infusion) | Arm E: JCAR017 Plus Relatlimab and/or Nivolumab (Post-JCAR017 Infusion) | Arm F: JCAR017 Plus CC-99282 (Post-JCAR017 Infusion)
Number analyzed (Participants) | 11 | 7 | 1 | 12 | 2 | 4
10^9 cells/L
  BASOPHILS (10^9/L) | 0.00 (0.009) | 0.03 (0.050) | 0.10 (NA) — Insufficient number of participants to calculate SD | -0.02 (0.038) | 0.05 (0.071) | 0.00 (0.075)
  EOSINOPHILS (10^9/L) | 0.20 (0.134) | 0.20 (0.282) | 0.00 (NA) — Insufficient number of participants to calculate SD | 0.01 (0.062) | -0.05 (0.071) | 0.04 (0.057)
  LYMPHOCYTES (10^9/L) | 0.40 (0.359) | 0.29 (0.138) | -0.60 (NA) — Insufficient number of participants to calculate SD | -0.20 (0.828) | 1.00 (0.707) | 0.87 (0.757)
  MONOCYTES (10^9/L) | 0.19 (0.209) | 0.38 (0.295) | 0.20 (NA) — Insufficient number of participants to calculate SD | -0.27 (0.527) | 0.15 (0.212) | 0.21 (0.279)
  NEUTROPHILS (10^9/L) | -1.69 (1.940) | -1.74 (1.312) | 2.30 (NA) — Insufficient number of participants to calculate SD | -4.98 (8.198) | 1.95 (3.889) | -2.47 (3.335)
  PLATELETS (10^9/L) | -6.91 (59.184) | 25.57 (28.547) | -77.00 (NA) — Insufficient number of participants to calculate SD | -125.92 (107.421) | -0.50 (20.506) | -11.00 (111.146)

8. Secondary Outcome: Change From Baseline in Percent of White Blood Cells
Description: Change from baseline in percent of white blood cells was measured using differential blood tests. A differential blood test is a blood test that measures the percentage and number of each type of white blood cell (WBC) - neutrophils, lymphocytes, monocytes, eosinophils and basophils - as well as abnormal cell types if they are present. These results are reported as percentages and absolute values, and compared against reference ranges to determine whether the values are normal, low, or high. Baseline is defined as the last measurement on or prior to any study treatment.
Time Frame: 85 days after the dose of JCAR017 for Arms A, B, D, E, and F; 57 days after the dose of JCAR017 for Arm C
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | Arm A: JCAR017 Plus Durvalumab (Post-JCAR017 Infusion) | Arm B: Cohort 1A | Arm C: JCAR017 Plus CC-220 (Iberdomide) (Post-JCAR017 Infusion) | Arm D: JCAR017 Plus Ibrutinib (Pre- and Post-JCAR017 Infusion) | Arm E: JCAR017 Plus Relatlimab and/or Nivolumab (Post-JCAR017 Infusion) | Arm F: JCAR017 Plus CC-99282 (Post-JCAR017 Infusion)
Number analyzed (Participants) | 11 | 7 | 1 | 12 | 2 | 4
Percent
  BASOPHILS/LEUKOCYTES (%) | 0.40 (0.420) | 0.89 (1.002) | 0.00 (NA) — Insufficient number of participants to calculate SD | 0.20 (0.558) | 0.15 (0.778) | 0.88 (1.450)
  EOSINOPHILS/LEUKOCYTES (%) | 1.24 (2.455) | 5.20 (6.491) | -1.00 (NA) — Insufficient number of participants to calculate SD | 1.02 (1.565) | -0.40 (0.283) | 1.45 (3.264)
  LYMPHOCYTES/LEUKOCYTES (%) | 11.59 (7.902) | 9.29 (4.870) | -37.00 (NA) — Insufficient number of participants to calculate SD | 2.60 (20.07) | 8.65 (1.202) | 24.73 (12.156)
  MONOCYTES/LEUKOCYTES (%) | 7.13 (3.955) | 11.43 (6.574) | -8.00 (NA) — Insufficient number of participants to calculate SD | 8.18 (14.077) | 1.30 (0.000) | 8.88 (2.724)
  NEUTROPHILS/LEUKOCYTES (%) | -20.69 (8.997) | -26.81 (13.462) | 45.00 (NA) — Insufficient number of participants to calculate SD | -12.13 (30.712) | -8.75 (0.354) | -35.55 (11.865)

9. Secondary Outcome: Change From Baseline Erythrocyte Numbers
Description: Change from baseline in erythrocyte (also known as red blood cell) numbers was measured using a test called a red blood cell count. Baseline is defined as the last measurement on or prior to any study treatment.
Time Frame: 85 days after the dose of JCAR017 for Arms A, B, D, E, and F; 57 days after the dose of JCAR017 for Arm C
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: 10^12 cells/L
Arm/Group | Arm A: JCAR017 Plus Durvalumab (Post-JCAR017 Infusion) | Arm B: Cohort 1A | Arm C: JCAR017 Plus CC-220 (Iberdomide) (Post-JCAR017 Infusion) | Arm D: JCAR017 Plus Ibrutinib (Pre- and Post-JCAR017 Infusion) | Arm E: JCAR017 Plus Relatlimab and/or Nivolumab (Post-JCAR017 Infusion) | Arm F: JCAR017 Plus CC-99282 (Post-JCAR017 Infusion)
Number analyzed (Participants) | 11 | 7 | 1 | 12 | 2 | 4
10^12 cells/L | -0.11 (0.507) | -0.21 (0.376) | -0.34 (NA) — Insufficient number of participants to calculate SD | -0.10 (0.476) | 0.05 (0.148) | -0.10 (0.281)

10. Secondary Outcome: Change From Baseline Hematocrit Ratio
Description: The change in the proportion of red blood cells in the blood was measured using a hematocrit test. A hematocrit test measures the volume of packed red blood cells relative to whole blood. This is represented as a ratio. Baseline is defined as the last measurement on or prior to any study treatment.
Time Frame: 85 days after the dose of JCAR017 for Arms A, B, D, E, and F; 57 days after the dose of JCAR017 for Arm C
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Arm A: JCAR017 Plus Durvalumab (Post-JCAR017 Infusion) | Arm B: Cohort 1A | Arm C: JCAR017 Plus CC-220 (Iberdomide) (Post-JCAR017 Infusion) | Arm D: JCAR017 Plus Ibrutinib (Pre- and Post-JCAR017 Infusion) | Arm E: JCAR017 Plus Relatlimab and/or Nivolumab (Post-JCAR017 Infusion) | Arm F: JCAR017 Plus CC-99282 (Post-JCAR017 Infusion)
Number analyzed (Participants) | 11 | 7 | 1 | 12 | 2 | 4
Ratio | 0.01 (0.048) | -0.02 (0.028) | -0.04 (NA) — Insufficient number of participants to calculate SD | 0.01 (0.048) | 0.02 (0.020) | -0.01 (0.039)

11. Secondary Outcome: Change From Baseline in Hemoglobin Levels
Description: The change from baseline in hemoglobin levels was measured using a hemoglobin test. A hemoglobin test measures the levels of hemoglobin in the blood. Hemoglobin is a protein in red blood cells that carries oxygen from the lungs to the rest of the body. Baseline is defined as the last measurement on or prior to any study treatment.
Time Frame: 85 days after the dose of JCAR017 for Arms A, B, D, E, and F; 57 days after the dose of JCAR017 for Arm C
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Arm A: JCAR017 Plus Durvalumab (Post-JCAR017 Infusion) | Arm B: Cohort 1A | Arm C: JCAR017 Plus CC-220 (Iberdomide) (Post-JCAR017 Infusion) | Arm D: JCAR017 Plus Ibrutinib (Pre- and Post-JCAR017 Infusion) | Arm E: JCAR017 Plus Relatlimab and/or Nivolumab (Post-JCAR017 Infusion) | Arm F: JCAR017 Plus CC-99282 (Post-JCAR017 Infusion)
Number analyzed (Participants) | 11 | 7 | 1 | 12 | 2 | 4
g/L | 0.45 (16.688) | -5.43 (12.869) | -12.00 (NA) — Insufficient number of participants to calculate SD | 1.38 (17.207) | 9.50 (13.435) | -2.50 (18.502)

12. Secondary Outcome: Change From Baseline in Specific Liver Serum Enzyme Levels
Description: Change from baseline in alanine aminotransferase (ALT) alkaline phosphatase (ALP), and aspartate aminotransferase (AST). Baseline is defined as the last measurement on or prior to any study treatment.
Time Frame: 85 days after the dose of JCAR017 for Arms A, B, D, E, and F; 57 days after the dose of JCAR017 for Arm C
Population: All treated participants with baseline and Day 85/Day 57 serum chemistry laboratory values. Prespecified to be reported per Arm and not per cohort.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Arm A: JCAR017 Plus Durvalumab (Post-JCAR017 Infusion) | Arm B: Cohort 1A | Arm C: JCAR017 Plus CC-220 (Iberdomide) (Post-JCAR017 Infusion) | Arm D: JCAR017 Plus Ibrutinib (Pre- and Post-JCAR017 Infusion) | Arm E: JCAR017 Plus Relatlimab and/or Nivolumab (Post-JCAR017 Infusion) | Arm F: JCAR017 Plus CC-99282 (Post-JCAR017 Infusion)
Number analyzed (Participants) | 11 | 7 | 1 | 12 | 2 | 4
U/L
  ALANINE AMINOTRANSFERASE (U/L) | 5.45 (5.429) | -2.86 (7.105) | -1.00 (NA) — Insufficient number of participants to calculate SD | -0.58 (11.237) | 0.50 (4.950) | 2.50 (2.082)
  ALKALINE PHOSPHATASE (U/L) | 12.09 (47.526) | -2.43 (24.234) | 22.00 (NA) — Insufficient number of participants to calculate SD | -18.50 (19.806) | 3.50 (16.263) | -16.25 (11.295)
  ASPARTATE AMINOTRANSFERASE (U/L) | 2.91 (5.467) | -4.43 (6.373) | -1.00 (NA) — Insufficient number of participants to calculate SD | 0.75 (7.008) | -5.50 (17.678) | -7.00 (7.439)

13. Secondary Outcome: Change From Baseline in Specific Serum Protein Levels
Description: Change from baseline in serum albumin and protein levels. Serum protein level tests are blood tests that measure the number of proteins in the blood. Baseline is defined as the last measurement on or prior to any study treatment.
Time Frame: 85 days after the dose of JCAR017 for Arms A, B, D, E, and F; 57 days after the dose of JCAR017 for Arm C
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Arm A: JCAR017 Plus Durvalumab (Post-JCAR017 Infusion) | Arm B: Cohort 1A | Arm C: JCAR017 Plus CC-220 (Iberdomide) (Post-JCAR017 Infusion) | Arm D: JCAR017 Plus Ibrutinib (Pre- and Post-JCAR017 Infusion) | Arm E: JCAR017 Plus Relatlimab and/or Nivolumab (Post-JCAR017 Infusion) | Arm F: JCAR017 Plus CC-99282 (Post-JCAR017 Infusion)
Number analyzed (Participants) | 11 | 7 | 1 | 12 | 2 | 4
g/L
  ALBUMIN (g/L) | 4.09 (5.281) | 2.29 (3.450) | 9.00 (NA) — Insufficient number of participants to calculate SD | 1.42 (4.926) | 6.00 (4.243) | 3.50 (9,747)
  PROTEIN (g/L) | 3.91 (8.166) | 0.00 (3.697) | 16.00 (NA) — Insufficient number of participants to calculate SD | -4.17 (3.881) | -0.50 (0.707) | -2.50 (11.030)

14. Secondary Outcome: Change From Baseline in Serum Beta-2-Microglobulin Levels
Description: Change from baseline in serum Beta-2-Microglobulin levels was measured using a beta-2 microglobulin (B2M) tumor marker test. Baseline is defined as the last measurement on or prior to any study treatment.
Time Frame: 85 days after the dose of JCAR017 for Arms A, B, D, E, and F; 57 days after the dose of JCAR017 for Arm C
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Arm A: JCAR017 Plus Durvalumab (Post-JCAR017 Infusion) | Arm B: Cohort 1A | Arm C: JCAR017 Plus CC-220 (Iberdomide) (Post-JCAR017 Infusion) | Arm D: JCAR017 Plus Ibrutinib (Pre- and Post-JCAR017 Infusion) | Arm E: JCAR017 Plus Relatlimab and/or Nivolumab (Post-JCAR017 Infusion) | Arm F: JCAR017 Plus CC-99282 (Post-JCAR017 Infusion)
Number analyzed (Participants) | 11 | 7 | 1 | 12 | 2 | 4
mg/L | 0.33 (0.735) | 0.06 (0.221) | -0.10 (NA) — Insufficient number of participants to calculate SD | -0.04 (1.019) | -0.65 (1.577) | 0.29 (0.654)

15. Secondary Outcome: Change From Baseline in Serum Bicarbonate Levels
Description: Change from baseline in serum bicarbonate levels was measured using a serum bicarbonate test. Baseline is defined as the last measurement on or prior to any study treatment.
Time Frame: 85 days after the dose of JCAR017 for Arms A, B, D, E, and F; 57 days after the dose of JCAR017 for Arm C
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Arm A: JCAR017 Plus Durvalumab (Post-JCAR017 Infusion) | Arm B: Cohort 1A | Arm C: JCAR017 Plus CC-220 (Iberdomide) (Post-JCAR017 Infusion) | Arm D: JCAR017 Plus Ibrutinib (Pre- and Post-JCAR017 Infusion) | Arm E: JCAR017 Plus Relatlimab and/or Nivolumab (Post-JCAR017 Infusion) | Arm F: JCAR017 Plus CC-99282 (Post-JCAR017 Infusion)
Number analyzed (Participants) | 11 | 7 | 1 | 12 | 2 | 4
mmol/L | 0.91 (3.270) | 0.00 (4.509) | 0.00 (NA) — Insufficient number of participants to calculate SD | -0.50 (4.079) | 3 (2.828) | -0.50 (2.646)

16. Secondary Outcome: Change From Baseline in Coagulation Times
Description: Change from baseline in activated partial thromboplastin and prothrombin times. Activated partial thromboplastin time and prothrombin time are blood tests that measure how long it takes for blood to form a clot. Baseline is defined as the last measurement on or prior to any study treatment.
Time Frame: 57 days after the dose of JCAR017
Population: All treated participants with baseline and Day 57 coagulation laboratory values. Prespecified to be reported per Arm and not per cohort.
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Arm A: JCAR017 Plus Durvalumab (Post-JCAR017 Infusion) | Arm B: Cohort 1A | Arm C: JCAR017 Plus CC-220 (Iberdomide) (Post-JCAR017 Infusion) | Arm D: JCAR017 Plus Ibrutinib (Pre- and Post-JCAR017 Infusion) | Arm E: JCAR017 Plus Relatlimab and/or Nivolumab (Post-JCAR017 Infusion) | Arm F: JCAR017 Plus CC-99282 (Post-JCAR017 Infusion)
Number analyzed (Participants) | 12 | 7 | 1 | 10 | 2 | 4
Seconds
  ACTIVATED PARTIAL THROMBOPLASTIN TIME (SEC) | -5.70 (21.348) | -0.31 (5.423) | 2.40 (NA) — Insufficient number of participants to calculate SD. | -2.25 (1.566) | 4.25 (6.859) | -2.10 (2.364)
  PROTHROMBIN TIME (SEC) | -0.02 (0.732) | 1.07 (2.974) | 0.40 (NA) — Insufficient number of participants to calculate SD. | -0.11 (0.479) | -2.90 (3.394) | 0.98 (2.695)

17. Secondary Outcome: Change From Baseline in D-Dimer Levels
Description: D-dimer is a substance that is produced in the body when blood clots are broken down. The D-dimer laboratory test measures the level of D-dimer in the blood and is often used to help diagnose or rule out conditions related to blood clotting, such as deep vein thrombosis (DVT) or pulmonary embolism (PE). Elevated levels of D-dimer may indicate the presence of a blood clot, but other factors can also cause an increase in D-dimer levels. Therefore, the D-dimer test is typically used in combination with other diagnostic tests to help make an accurate diagnosis. Baseline is defined as the last measurement on or prior to any study treatment.
Time Frame: 57 days after the dose of JCAR017
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Arm A: JCAR017 Plus Durvalumab (Post-JCAR017 Infusion) | Arm B: Cohort 1A | Arm C: JCAR017 Plus CC-220 (Iberdomide) (Post-JCAR017 Infusion) | Arm D: JCAR017 Plus Ibrutinib (Pre- and Post-JCAR017 Infusion) | Arm E: JCAR017 Plus Relatlimab and/or Nivolumab (Post-JCAR017 Infusion) | Arm F: JCAR017 Plus CC-99282 (Post-JCAR017 Infusion)
Number analyzed (Participants) | 12 | 7 | 1 | 10 | 2 | 4
mg/L | -0.92 (1.789) | -0.13 (0.311) | -0.46 (NA) — Insufficient number of participants to calculate SD. | -0.69 (1.601) | -0.39 (0.746) | 0.13 (0.241)

18. Secondary Outcome: Change From Baseline in Fibrinogen Levels
Description: Fibrinogen is a protein that plays a role in a number of processes in the body, including blood clot formation, wound healing, inflammation, and blood vessel growth. Baseline is defined as the last measurement on or prior to any study treatment.
Time Frame: 57 days after the dose of JCAR017
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Arm A: JCAR017 Plus Durvalumab (Post-JCAR017 Infusion) | Arm B: Cohort 1A | Arm C: JCAR017 Plus CC-220 (Iberdomide) (Post-JCAR017 Infusion) | Arm D: JCAR017 Plus Ibrutinib (Pre- and Post-JCAR017 Infusion) | Arm E: JCAR017 Plus Relatlimab and/or Nivolumab (Post-JCAR017 Infusion) | Arm F: JCAR017 Plus CC-99282 (Post-JCAR017 Infusion)
Number analyzed (Participants) | 12 | 7 | 1 | 10 | 2 | 4
g/L | -0.23 (1.379) | -0.65 (1.697) | 2.59 (NA) — Insufficient number of participants to calculate SD. | -2.04 (2.012) | -5.12 (1.888) | -1.77 (0.525)

19. Secondary Outcome: Change From Baseline in Prothrombin International Normalized Ratio
Description: The Prothrombin International Normalized Ratio (INR) is used to determine the clotting tendency of blood. The INR is derived from prothrombin time (PT) which is calculated as a ratio of the patient's PT to a control PT. Baseline is defined as the last measurement on or prior to any study treatment.
Time Frame: 57 days after the dose of JCAR017
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Arm A: JCAR017 Plus Durvalumab (Post-JCAR017 Infusion) | Arm B: Cohort 1A | Arm C: JCAR017 Plus CC-220 (Iberdomide) (Post-JCAR017 Infusion) | Arm D: JCAR017 Plus Ibrutinib (Pre- and Post-JCAR017 Infusion) | Arm E: JCAR017 Plus Relatlimab and/or Nivolumab (Post-JCAR017 Infusion) | Arm F: JCAR017 Plus CC-99282 (Post-JCAR017 Infusion)
Number analyzed (Participants) | 12 | 7 | 1 | 10 | 2 | 4
Ratio | -0.01 (0.079) | 0.08 (0.234) | 0.10 (NA) — Insufficient number of participants to calculate SD. | -0.01 (0.066) | -0.20 (0.283) | 0.10 (0.198)

20. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS is defined as time from JCAR017 infusion to disease progression or death from any cause.
  Progressive disease (PD) was measured using CT and PET as an increase in size index and non-index lesions, spleen size, and the presence of new lesions or diseased bone marrow.
  Summarized using Kaplan-Meier estimates.
Time Frame: From JCAR017 infusion to disease progression or death from any cause (up to approximately 62 months)
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A: JCAR017 Plus Durvalumab (Post-JCAR017 Infusion) | Arm B: Cohort 1A | Arm C: JCAR017 Plus CC-220 (Iberdomide) (Post-JCAR017 Infusion) | Arm D: JCAR017 Plus Ibrutinib (Pre- and Post-JCAR017 Infusion) | Arm E: JCAR017 Plus Relatlimab and/or Nivolumab (Post-JCAR017 Infusion) | Arm F: JCAR017 Plus CC-99282 (Post-JCAR017 Infusion)
Number analyzed (Participants) | 14 | 8 | 1 | 15 | 2 | 5
Months | 20.90 [2.96 to NA] — Upper CI could not be calculated due to insufficient number of events. | NA [2.30 to NA] — PFS could not be calculated due to insufficient number of events. | 2.86 [NA to NA] — Upper and lower CI could not be calculated due to insufficient number of events. | NA [1.91 to NA] — PFS could not be calculated due to insufficient number of events. | 4.07 [2.17 to NA] — Upper CI could not be calculated due to insufficient number of events. | 3.06 [2.79 to NA] — Upper CI could not be calculated due to insufficient number of events.

21. Secondary Outcome: Overall Survival (OS)
Description: Time from JCAR017 infusion to death. Data from surviving participants was censored at the last time that the participant was known to be alive.
  Summarized using Kaplan-Meier estimates.
Time Frame: From start of JCAR017 to time of death from any cause, or data cut-off date, whichever occurred first (up to approximately 62 months)
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A: JCAR017 Plus Durvalumab (Post-JCAR017 Infusion) | Arm B: Cohort 1A | Arm C: JCAR017 Plus CC-220 (Iberdomide) (Post-JCAR017 Infusion) | Arm D: JCAR017 Plus Ibrutinib (Pre- and Post-JCAR017 Infusion) | Arm E: JCAR017 Plus Relatlimab and/or Nivolumab (Post-JCAR017 Infusion) | Arm F: JCAR017 Plus CC-99282 (Post-JCAR017 Infusion)
Number analyzed (Participants) | 14 | 8 | 1 | 15 | 2 | 5
Months | 31.34 [4.50 to 38.08] | NA [3.22 to NA] — Insufficient number of events to calculate Median OS and upper CI limit. | 2.86 [NA to NA] — Insufficient participants calculate lower and upper CI limits. | NA [9.46 to NA] — Insufficient number of events to calculate Median OS and upper CI limit. | NA [7.26 to NA] — Insufficient number of events to calculate Median OS and upper CI limit. | 6.60 [4.27 to NA] — Insufficient number of events to calculate upper CI limit.

22. Secondary Outcome: Overall Response Rate (ORR)
Description: The ORR is the percent of participants achieving an objective response of partial response (PR) or better according to the Lugano Criteria for Response Assessment (Cheson, 2014), prior to start of another non-study anticancer therapy.
  Complete response (CR) assessed by CT-scan:
  * Index lesions: Nodal Disease: ≤ 1.5 cm in largest transverse diameter, Extranodal Disease: Absent
  * Non-index lesions: Absent,
  * Spleen: <13 cm
  * New lesions: None
  * Bone marrow: Normal
  Partial response (PR) assessed by CT-scan:
  * Index lesions: >=50% decrease from baseline in shortest diameter
  * Non-index lesions: No increase,
  * Spleen: >50% decrease from baseline in enlarged portion
  * New lesions: None
  * Bone marrow: N/A Overall Response (OR) = CR + PR
Time Frame: At 1, 3, 6, 9, 12, 18 and 24 months post-JCAR017 infusion
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percent of Participants
Arm/Group | Arm A: JCAR017 Plus Durvalumab (Post-JCAR017 Infusion) | Arm B: Cohort 1A | Arm C: JCAR017 Plus CC-220 (Iberdomide) (Post-JCAR017 Infusion) | Arm D: JCAR017 Plus Ibrutinib (Pre- and Post-JCAR017 Infusion) | Arm E: JCAR017 Plus Relatlimab and/or Nivolumab (Post-JCAR017 Infusion) | Arm F: JCAR017 Plus CC-99282 (Post-JCAR017 Infusion)
Number analyzed (Participants) | 14 | 8 | 1 | 15 | 2 | 5
Percent of Participants
  Month 1 | 92.9 [66.1 to 99.8] | 75.0 [34.9 to 96.8] | 100.0 [2.5 to 100.0] | 60.0 [32.3 to 83.7] | 100.00 [15.8 to 100.0] | 60.0 [14.7 to 94.7]
  Month 3 | 92.9 [66.1 to 99.8] | 75.0 [34.9 to 96.8] | 100.0 [2.5 to 100.0] | 73.3 [44.9 to 92.2] | 100.0 [15.8 to 100.0] | 60.0 [14.7 to 94.7]
  Month 6 | 92.9 [66.1 to 99.8] | 75.0 [34.9 to 96.8] | 100.0 [2.5 to 100.0] | 73.3 [44.9 to 92.2] | 100.0 [15.8 to 100.0] | 60.0 [14.7 to 94.7]
  Month 9 | 92.9 [66.1 to 99.8] | 75.0 [34.9 to 96.8] | 100.0 [2.5 to 100.0] | 73.3 [44.9 to 92.2] | 100.0 [15.8 to 100.0] | 60.0 [14.7 to 94.7]
  Month 12 | 92.9 [66.1 to 99.8] | 75.0 [34.9 to 96.8] | 100.0 [2.5 to 100.0] | 73.3 [44.9 to 92.2] | 100.0 [15.8 to 100.0] | 60.0 [14.7 to 94.7]
  Month 18 | 92.9 [66.1 to 99.8] | 75.0 [34.9 to 96.8] | 100.0 [2.5 to 100.0] | 73.3 [44.9 to 92.2] | 100.0 [15.8 to 100.0] | 60.0 [14.7 to 94.7]
  Month 24 | 92.9 [66.1 to 99.8] | 75.0 [34.9 to 96.8] | 100.0 [2.5 to 100.0] | 73.3 [44.9 to 92.2] | 100.0 [15.8 to 100.0] | 60.0 [14.7 to 94.7]

23. Secondary Outcome: Duration of Response (DOR)
Description: DOR is defined as the time from first response to disease progression or death from any cause.
  Summarized using Kaplan-Meier estimates.
Time Frame: From JCAR017 infusion to disease progression or death from any cause (up to approximately 62 months)
Population: All Responders in Combination Treated Set. The combination treated set included all participants who received an infusion of conforming JCAR017 cell product and at least one dose of the combination agent. Prespecified to be reported per Arm and not per cohort.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A: JCAR017 Plus Durvalumab (Post-JCAR017 Infusion) | Arm B: Cohort 1A | Arm C: JCAR017 Plus CC-220 (Iberdomide) (Post-JCAR017 Infusion) | Arm D: JCAR017 Plus Ibrutinib (Pre- and Post-JCAR017 Infusion) | Arm E: JCAR017 Plus Relatlimab and/or Nivolumab (Post-JCAR017 Infusion) | Arm F: JCAR017 Plus CC-99282 (Post-JCAR017 Infusion)
Number analyzed (Participants) | 13 | 6 | 1 | 11 | 2 | 3
Months | 21.45 [2.43 to NA] — Insufficient number of events to calculate upper CI limit. | NA [1.45 to NA] — Insufficient number of events to calculate DoR and upper CI limit. | 1.91 [NA to NA] — Insufficient number of participants to calculate upper and lower CI limits. | NA [17.71 to NA] — Insufficient number of events to calculate DoR upper CI limit. | 3.15 [1.22 to NA] — Insufficient number of events to calculate upper CI limit. | 3.29 [1.87 to NA] — Insufficient number of events to calculate upper CI limit

24. Secondary Outcome: Event-Free Survival (EFS)
Description: EFS is defined as time from JCAR017 infusion to disease progression, starting a new antilymphoma therapy, or death from any cause, whichever occurred first.
Time Frame: From JCAR017 infusion to disease progression or death from any cause (up to approximately 62 months)
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A: JCAR017 Plus Durvalumab (Post-JCAR017 Infusion) | Arm B: Cohort 1A | Arm C: JCAR017 Plus CC-220 (Iberdomide) (Post-JCAR017 Infusion) | Arm D: JCAR017 Plus Ibrutinib (Pre- and Post-JCAR017 Infusion) | Arm E: JCAR017 Plus Relatlimab and/or Nivolumab (Post-JCAR017 Infusion) | Arm F: JCAR017 Plus CC-99282 (Post-JCAR017 Infusion)
Number analyzed (Participants) | 14 | 8 | 1 | 15 | 2 | 5
Months | 20.90 [2.96 to NA] — Insufficient number of events to calculate upper CI limit. | NA [2.30 to NA] — Insufficient number of events to calculate EFS and upper CI limit. | 2.86 [NA to NA] — Insufficient number of participants to calculate lower and upper CI limits. | 18.76 [1.91 to NA] — Insufficient number of events to calculate upper CI limit. | 4.07 [2.17 to NA] — Insufficient number of events to calculate upper CI limit. | 3.06 [2.79 to NA] — Insufficient number of events to calculate upper CI limit.

25. Secondary Outcome: Maximum Concentration (Cmax) of JCAR017 by qPCR
Description: Cmax is the maximum or peak concentration of drug reached in the plasma following a dose of the drug.
  qPCR was used to determine Cmax by detecting the JCAR017 transgene.
Time Frame: Up to 24 months post- JCAR017 infusion
Population: All participants who received an infusion of conforming JCAR017 cell product with baseline and on-study PK measurements. Prespecified to be reported per Arm and not per cohort.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Copies/ug
Arm/Group | Arm A: JCAR017 Plus Durvalumab (Post-JCAR017 Infusion) | Arm B: Cohort 1A | Arm C: JCAR017 Plus CC-220 (Iberdomide) (Post-JCAR017 Infusion) | Arm D: JCAR017 Plus Ibrutinib (Pre- and Post-JCAR017 Infusion) | Arm E: JCAR017 Plus Relatlimab and/or Nivolumab (Post-JCAR017 Infusion) | Arm F: JCAR017 Plus CC-99282 (Post-JCAR017 Infusion)
Number analyzed (Participants) | 15 | 10 | 1 | 13 | 2 | 5
Copies/ug | 11464.7 (305.8) | 14087.1 (434.7) | 28845.0 (NA) — Insufficient number of participants to calculate geometric CV. | 28877.7 (314.2) | 58522.9 (63.5) | 18003.4 (343.4)

26. Secondary Outcome: Time to Maximum Concentration (Tmax) of JCAR017 by qPCR
Description: Time to maximum concentration (Tmax) is the time it takes for a drug to reach the maximum concentration (Cmax) after administration.
  qPCR was used to determine Tmax by detecting the JCAR017 transgene.
Time Frame: Up to 24 months post- JCAR017 infusion
Population: All participants who received an infusion of conforming JCAR017 cell product (JCAR017 PK analysis) or at least 1 dose of combination agent (combination agent analysis) with baseline and on-study PK measurements. Prespecified to be reported per Arm and not per cohort.
Measure: Median (Full Range); unit: Days
Arm/Group | Arm A: JCAR017 Plus Durvalumab (Post-JCAR017 Infusion) | Arm B: Cohort 1A | Arm C: JCAR017 Plus CC-220 (Iberdomide) (Post-JCAR017 Infusion) | Arm D: JCAR017 Plus Ibrutinib (Pre- and Post-JCAR017 Infusion) | Arm E: JCAR017 Plus Relatlimab and/or Nivolumab (Post-JCAR017 Infusion) | Arm F: JCAR017 Plus CC-99282 (Post-JCAR017 Infusion)
Number analyzed (Participants) | 15 | 10 | 1 | 13 | 2 | 5
Days | 10.0 [7.0 to 42.0] | 10.0 [7.0 to 19.0] | 29.0 [29.0 to 29.0] | 14.0 [7.0 to 28.0] | 10.0 [10.0 to 10.0] | 8.5 [7.0 to 10.0]

27. Secondary Outcome: Total Exposure to JCAR017 as Measured by the Area Under the Curve (AUC) by qPCR
Description: Area Under the Curve" (AUC) represents the total exposure of participants to study drug. qPCR was used to determine AUC by detecting the JCAR017 transgene.
Time Frame: Up to 24 months post- JCAR017 infusion
Population: as for outcome 25
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Copies/ug*day
Arm/Group | Arm A: JCAR017 Plus Durvalumab (Post-JCAR017 Infusion) | Arm B: Cohort 1A | Arm C: JCAR017 Plus CC-220 (Iberdomide) (Post-JCAR017 Infusion) | Arm D: JCAR017 Plus Ibrutinib (Pre- and Post-JCAR017 Infusion) | Arm E: JCAR017 Plus Relatlimab and/or Nivolumab (Post-JCAR017 Infusion) | Arm F: JCAR017 Plus CC-99282 (Post-JCAR017 Infusion)
Number analyzed (Participants) | 15 | 10 | 1 | 13 | 2 | 5
Copies/ug*day | 85169.458 (237.850) | 83155.476 (473.149) | 288951.250 (NA) — Insufficient number of participants to calculate geometric CV. | 281265.838 (360.545) | 529755.009 (9.534) | 190904.832 (224.399)

ADVERSE EVENTS:
Time Frame: Participants were assessed for All-Cause Mortality from the date of leukapheresis until study completion (assessed up to approximately 62 months). SAEs and Other AEs were assessed from leukapheresis to 90 days after last dose of study therapy (an average of 7.5 months up until a max of 10.5 months).
Description: All-Cause Mortality, Serious Adverse Events and Other (Not Including Serious) Adverse Events represents all participants that underwent leukapheresis and may or may not have received at least 1 dose of JCAR017. Data is shown per cohort.
Arm/Group | Arm A: Cohort 1A JCAR017 Plus Durvalumab (Post-JCAR017 Infusion) | Arm A: Cohort 1B JCAR017 Plus Durvalumab (Post-JCAR017 Infusion) | Arm B: Cohort 1A JCAR017 Plus CC-122 (Post-JCAR017 Infusion) | Arm C: Cohort 1A JCAR017 Plus CC-220 (Iberdomide) (Post-JCAR017 Infusion) | Arm D: Cohort 1A JCAR017 Plus Ibrutinib (Pre- and Post-JCAR017 Infusion) | Arm E: Cohort 1C JCAR017 Plus Relatlimab and/or Nivolumab (Post-JCAR017 Infusion) | Arm F: Cohort 1A Cohort 1A and 1D JCAR017 Plus CC-99282 (Post-JCAR017 Infusion) | Arm F: Cohort 1D Cohort 1A and 1D JCAR017 Plus CC-99282 (Post-JCAR017 Infusion)
All-Cause Mortality (participants affected / at risk) | 7/11 | 7/9 | 8/13 | 1/1 | 5/17 | 1/2 | 4/7 | 1/2
Serious Adverse Events (participants affected / at risk) | 4/11 | 6/9 | 7/13 | 1/1 | 6/17 | 2/2 | 3/7 | 0/2
Other Adverse Events (participants affected / at risk) | 8/11 | 8/9 | 11/13 | 1/1 | 17/17 | 2/2 | 4/7 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Cohort 1A JCAR017 Plus Durvalumab (Post-JCAR017 Infusion) (N=11) | Arm A: Cohort 1B JCAR017 Plus Durvalumab (Post-JCAR017 Infusion) (N=9) | Arm B: Cohort 1A JCAR017 Plus CC-122 (Post-JCAR017 Infusion) (N=13) | Arm C: Cohort 1A JCAR017 Plus CC-220 (Iberdomide) (Post-JCAR017 Infusion) (N=1) | Arm D: Cohort 1A JCAR017 Plus Ibrutinib (Pre- and Post-JCAR017 Infusion) (N=17) | Arm E: Cohort 1C JCAR017 Plus Relatlimab and/or Nivolumab (Post-JCAR017 Infusion) (N=2) | Arm F: Cohort 1A Cohort 1A and 1D JCAR017 Plus CC-99282 (Post-JCAR017 Infusion) (N=7) | Arm F: Cohort 1D Cohort 1A and 1D JCAR017 Plus CC-99282 (Post-JCAR017 Infusion) (N=2)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Arrhythmia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Colitis ischaemic (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Enteritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Cytokine release syndrome (Immune system disorders) | 0 | 1 | 3 | 0 | 0 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0
Respiratory syncytial virus infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Staphylococcal sepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypervolaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Colon cancer stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Agraphia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Encephalopathy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Neurotoxicity (Nervous system disorders) | 1 | 1 | 2 | 0 | 2 | 1 | 1 | 0
Mental status changes (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Large intestine perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Cohort 1A JCAR017 Plus Durvalumab (Post-JCAR017 Infusion) (N=11) | Arm A: Cohort 1B JCAR017 Plus Durvalumab (Post-JCAR017 Infusion) (N=9) | Arm B: Cohort 1A JCAR017 Plus CC-122 (Post-JCAR017 Infusion) (N=13) | Arm C: Cohort 1A JCAR017 Plus CC-220 (Iberdomide) (Post-JCAR017 Infusion) (N=1) | Arm D: Cohort 1A JCAR017 Plus Ibrutinib (Pre- and Post-JCAR017 Infusion) (N=17) | Arm E: Cohort 1C JCAR017 Plus Relatlimab and/or Nivolumab (Post-JCAR017 Infusion) (N=2) | Arm F: Cohort 1A Cohort 1A and 1D JCAR017 Plus CC-99282 (Post-JCAR017 Infusion) (N=7) | Arm F: Cohort 1D Cohort 1A and 1D JCAR017 Plus CC-99282 (Post-JCAR017 Infusion) (N=2)
Anaemia (Blood and lymphatic system disorders) | 3 | 7 | 5 | 1 | 10 | 2 | 2 | 1
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypofibrinogenaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 3 | 3 | 4 | 0 | 0 | 1 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 1 | 1 | 3 | 0 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 2 | 5 | 8 | 1 | 5 | 2 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 4 | 4 | 7 | 1 | 2 | 2 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Extrasystoles (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0
Supraventricular extrasystoles (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Cerumen impaction (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Dry eye (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Eye irritation (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Periorbital oedema (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Visual impairment (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vitreous floaters (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 1 | 1 | 1 | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Anal incontinence (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Chapped lips (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 3 | 3 | 1 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 3 | 0 | 3 | 1 | 1 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Enterocolitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hiatus hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ileus paralytic (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mesenteric artery stenosis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 4 | 2 | 5 | 1 | 0 | 0 | 0 | 1
Oral pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Proctalgia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 4 | 0 | 2 | 0 | 3 | 0 | 0 | 0
Asthenia (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chills (General disorders) | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 0
Fatigue (General disorders) | 3 | 4 | 6 | 0 | 2 | 0 | 0 | 2
Mucosal inflammation (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oedema (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 1
Pain (General disorders) | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 0
Physical deconditioning (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 2 | 0 | 1 | 2 | 0 | 0 | 1
Suprapubic pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Swelling (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Jaundice (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ocular icterus (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cytokine release syndrome (Immune system disorders) | 0 | 3 | 2 | 1 | 7 | 2 | 1 | 1
Hypogammaglobulinaemia (Immune system disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Candida infection (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cytomegalovirus infection reactivation (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 2 | 0 | 1 | 0 | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Viral infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vulvitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0 | 2 | 1 | 0 | 0
Epicondylitis (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vascular access site bruising (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Blood uric acid increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
International normalised ratio increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Liver function test increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 0 | 10 | 0 | 1 | 1
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 0 | 11 | 0 | 3 | 2
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 9 | 0 | 1 | 2
Prostatic specific antigen increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 12 | 0 | 2 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 2 | 3 | 1 | 5 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 2 | 1 | 1 | 2 | 1 | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 | 4 | 1 | 0 | 2 | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 3 | 3 | 1 | 1 | 1 | 0 | 0
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 3 | 1 | 1 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 4 | 1 | 0 | 0 | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1
Coccydynia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Mastication disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2 | 0 | 3 | 1 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Colorectal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Amnesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Brain fog (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 5 | 1 | 3 | 0 | 1 | 0
Dysarthria (Nervous system disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyporeflexia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypotonia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Intention tremor (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Memory impairment (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Neuralgia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Neurotoxicity (Nervous system disorders) | 0 | 1 | 2 | 1 | 3 | 1 | 0 | 0
Nystagmus (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Peripheral motor neuropathy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Peroneal nerve palsy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Resting tremor (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Restless legs syndrome (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tremor (Nervous system disorders) | 0 | 1 | 2 | 0 | 2 | 0 | 0 | 1
Agitation (Psychiatric disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 0
Delirium (Psychiatric disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Depressed mood (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 2 | 0 | 0 | 0 | 3 | 0 | 0 | 1
Libido decreased (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Chronic kidney disease (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Micturition urgency (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Urinary tract pain (Renal and urinary disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Urine abnormality (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 2 | 0 | 1 | 1 | 1 | 0
Diaphragmalgia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 2 | 0 | 1 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 2 | 0 | 0 | 0
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 3 | 0 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 1 | 2 | 0 | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Aneurysm (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bloody discharge (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Embolism (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Flushing (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0 | 0 | 3 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 2 | 2 | 1 | 1 | 0 | 0 | 2
Orthostatic hypotension (Vascular disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Appetite disorder (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Thrombophlebitis (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-01-27): https://cdn.clinicaltrials.gov/large-docs/19/NCT03310619/Prot_SAP_000.pdf